CLINICAL TRIAL: NCT06387316
Title: Cephalic Phase Responses to Nutritive and Non-Nutritive Sweeteners
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2023-1526
Record Dates: First submitted 2024-03-27; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Pre Diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Masking Description: solutions are coded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- No Oral Stimulation (Other): No oral stimulation is provided.
  Interventions: Other: No Oral Stimulation
- Oral Water Stimulation (Other): Oral stimulation with water.
  Interventions: Other: Oral water stimulation
- Oral Salt Stimulation (Other): Oral stimulation with salt.
  Interventions: Other: Oral Salt Stimulation
- Oral Sucralose Stimulation (Other): Oral stimulation with sucralose.
  Interventions: Other: Oral Sucralose Stimulation
- Oral Sucrose stimulation (Other): Oral stimulation with sucrose.
  Interventions: Other: No Oral Stimulation; Other: Oral Sucrose stimulation

INTERVENTIONS:
Other: No Oral Stimulation — No oral stimulation
  Arms: No Oral Stimulation; Oral Sucrose stimulation
Other: Oral water stimulation — Oral water stimulation
  Arms: Oral Water Stimulation
Other: Oral Salt Stimulation — Oral Salt Stimulation
  Arms: Oral Salt Stimulation
Other: Oral Sucralose Stimulation — Oral Sucralose Stimulation
  Arms: Oral Sucralose Stimulation
Other: Oral Sucrose stimulation — Oral Sucrose stimulation
  Arms: Oral Sucrose stimulation

SUMMARY:
This study will focus on changes in blood sugar in response to tasting different types of sweeteners using continuous glucose monitoring (CGM) technology.

DETAILED DESCRIPTION:
Participants will be recruited through posting of advertisements about the study. Flyers will be posted on and off campus. Individuals interested in the study will contact the researchers and an initial appointment will be scheduled.

First Lab Visit (Day 1):

Consent and Instruction: Researchers will explain the study procedures, including the use of continuous glucose monitoring (CGM), home-based taste testing and wearing the Fitbit activity tracker. Participants will complete a short questionnaire (screening questionnaire) that elicits demographic, health and activity information. Participants can choose to decline to answer any questions they prefer not to answer. Researchers will determine if participants meet eligibility criteria and participants will then decide if they want to participate. A CGM device will be placed on the participant's arm to monitor glucose levels continuously. Placing the monitor involves putting an egg-shaped plastic container (about the size of a golf ball) on the back of one arm and a button is pushed and this presses the sensor on the arm. It is held on by adhesive. It is like applying a band aid though there is a hair-like flexible fiber that is pressed into the skin (not into a vein). The participant feels little more than mild pressure - far less than a needle stick. Participants will be given individually portioned, labeled sample solutions including a nutritive sweetener, non-nutritive sweetener, a non-sweet control stimulus (salt) and just water along with commercially available no sodium rice cakes (cut to bite-size pieces). Participants will be instructed to place one rice cake sample in their mouth and sip a 5ml oral solution sample and masticate for 15 seconds and expectorate. This will be repeated 3 additional times. With about 15 seconds between samples. This exposure will require about 2 minutes. This will be repeated 4 times a day (before breakfast, before lunch, before dinner and at 8PM) on 8 days. There will be no oral stimulation for 2 days. Participants will be provided with activity recall sheets and instructed to record their sleep patterns, and physical activity for 10 days. This form will only contain an identification code, no personally identifiable information be on the form. Participants will also be asked to wear a Fitbit to monitor activity. This is exactly like wearing a wristwatch.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 to 70 years old will be eligible to participate.
* Good health and without known medical conditions, including but not limited to, diabetes, cardiovascular diseases, metabolic disorders, and any other chronic conditions that could significantly affect glycemia.
* No history of major surgeries, organ transplantations, or significant medical interventions that might impact glycemia.
* No medications that could interfere with glucose metabolism or sweet taste perception. Use of vitamins or contraceptives will be permissible if continued for the 12 days of study participation.
* No dietary restrictions or sensitivities that prevent them from tasting or swishing sweeteners and rice cakes provided during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Blood glucose concentration | 10 days
  blood glucose concentration measured by continuous glucose monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No